CLINICAL TRIAL: NCT05559086
Title: Neutrophils to Lymphocytes and Platelets Ratio (N/LP) as Predictor of Mortality in Septic- Acute Kidney Injury Patients
Brief Title: N/LP Ratio as Predictor of Mortality in Septic AKI Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Kamel Mohamed Abd elhaq (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Kamel Mohamed Abd elhaq, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: N/LP in septic AKI
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury Due to Sepsis
Keywords: Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the role of Neutrophils to lymphocytes and platelets ratio (N/LP ratio) as a biomarkers for mortality in septic -AKI

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a rapid deteriorattion in renal function,and AKI is frequent in hospitalized patients and its incidence is higher in critically ill patients, in whom the leading cause of AKI is sepsis,.Sepsis is the systemic inflammatory response to an infectious insult, . Septic-AKI patients have higher severity scores at admission, more non-renal organ failure and requirement of vasopressors and mechanical ventilation.

AKI has been associated with longer hospital stays, in-hospital mortality, progression to chronic kidney disease . Septic-AKI also has higher short-term mortality rate, prolonged length of hospital stays and higher probability of renal function recovery at hospital discharge.Therefore, it is important to detect predictors of AKI and mortality to prevent, diagnose and treat this complication..

A recent study demonstrated that septic AKI patients have higher detectable plasma and urine neutrophil gelatinase associated lipocalin (NGAL) compared with nonseptic AKI patients.The utility of these and other novel biomarkers including cystatin C, liver fatty acid-binding protein (L-FABP), and netrin-1 for early detection of sepsis-induced AKI is very encouraging and may have prognostic as well as pathogenetic implications. For instance, urinary liver fatty acid-binding protein (L-FABP) is significantly higher in AKI than non-AKI in adult ICU patients. On the other hand, netrin-1, is excreted in the urine as early as 1 hour after injury reaching approximately 30-fold increase by 3 hours . The utility of such biomarkers may be of particular importance because early detection of AKI will allow for appropriate and timely interventions that would significantly decrease morbidity and mortality related to AKI.

Recent studies have shown that the level of urinary biomarkers like interleukin-18 (IL-8), neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule-1 (KIM-1) increases in the early stage of AKI, prior to creatinine elevation and histological changes, which may contribute to the early detection of AKI. these are sensitive and specific biomarkers for the early diagnosis of AKI in septic patients

Indeed, the role of intrarenal and systemic inflammation appears to be significant in the pathophysiology of septic-AKI and in the associated multi-organ dysfunction

For septic AKI treatment options are limited, and mortality remains high.

The neutrophil to lymphocyte ratio (N/L ratio) and neutrophil to lymphocytes and platelets ratio (N/LP ratio) have been associated with AKI in the emergency setting ,sepsis, contrast induced-AKI, cardiovascular surgery and abdominal surgery. These are easily calculated, effective , and inexpensive markers of systemic inflammation which might be promising in AKI patients. The NL ratio was a predictive of mortality thus, platelet count was incorporated in the ratio to increase its sensitivity in predicting patient outcomes as In the early phases of sepsis platelet/neutrophils complexes are raised, and reduced in severe and complicated sepsis due to peripheral sequestration or sepsis-associated thrombocytopenia.

The prognostic ability of the neutrophils to lymphocytes and platelets ratio (N/LP ratio) has not previously been evaluated in septic-AKI. the N/LP ratio at admission was an independent predictor of mortality in patients who develop septic-AKI within the first week of admission. More importantly, a N/LP ratio lower than 14 is predictive of patient survival, which further reflects that lower inflammation is associated with lower mortality in critically ill septic patients and a higher N/LP ratio at ICU admission was independently associated with in-hospital mortality in septic-AKI patients Thus, highlighting the role of the N/LP ratio as a significant marker of systemic inflammatory response at ICU admission.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and older
2. Diagnosed as Septic -AKI

   AKI was diagnosed according to kdigo definition and staging

   Sepsis was diagnosed according to the third international consensus definitions as an acute change in total Sequential Organ Failure Assessment (SOFA) score ≥2 points consequent to the infection.
3. CRP as marker of sepsis
4. CBC as marker of sepsis, N/LP ratio is calculated as: (Neutrophil count × 100)/(Lymphocyte count × Platelet count). the N/LP ratio lower than 14 is predictive of patient survival, which further reflects that lower inflammation is associated with lower mortality in critically ill septic patients. Thus, highlighting the role of the N/LP ratio as a significant marker of systemic inflammatory response at ICU admission.

Exclusion Criteria:

* 1.prerenal and post renal AKI

  2.Contrast induced AKI

  3. Drugs induced AKI

  4.CKD patients and ESRD patient

  5.Active Lupus, LN

  6.Malignancies

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and older
  Diagnosed as AKI due to sepsis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-25 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Neutrophils to Lymphocytes and platelets ratio (N/LP) as predictor of mortality in septic- acute kidney injury patients | Baseline
  The N/LP ratio at icu admission was independently associated with in-hospital mortality in septic-AKI patients the assessment of this ratio is straight forward from routine blood analysis in ICU patients useful in identifying patients at risk of mortality The N/LP ratio at icu admission was independently associated with in-hospital mortality in septic-AKI patients the assessment of this ratio is straight forward from routine blood analysis in ICU patients useful in identifying patients at risk of mortality

REFERENCES:
- [Background] Kellum JA, Prowle JR. Paradigms of acute kidney injury in the intensive care setting. Nat Rev Nephrol. 2018 Apr;14(4):217-230. doi: 10.1038/nrneph.2017.184. Epub 2018 Jan 22. PMID 29355173
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Nguyen HB, Smith D. Sepsis in the 21st century: recent definitions and therapeutic advances. Am J Emerg Med. 2007 Jun;25(5):564-71. doi: 10.1016/j.ajem.2006.08.015. PMID 17543662
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Zarjou A, Agarwal A. Sepsis and acute kidney injury. J Am Soc Nephrol. 2011 Jun;22(6):999-1006. doi: 10.1681/ASN.2010050484. Epub 2011 May 12. PMID 21566052
- [Background] Prowle JR, Bellomo R. Sepsis-associated acute kidney injury: macrohemodynamic and microhemodynamic alterations in the renal circulation. Semin Nephrol. 2015 Jan;35(1):64-74. doi: 10.1016/j.semnephrol.2015.01.007. PMID 25795500
- [Background] Gomez H, Ince C, De Backer D, Pickkers P, Payen D, Hotchkiss J, Kellum JA. A unified theory of sepsis-induced acute kidney injury: inflammation, microcirculatory dysfunction, bioenergetics, and the tubular cell adaptation to injury. Shock. 2014 Jan;41(1):3-11. doi: 10.1097/SHK.0000000000000052. PMID 24346647
- [Background] Martensson J, Bellomo R. Pathophysiology of Septic Acute Kidney Injury. Contrib Nephrol. 2016;187:36-46. doi: 10.1159/000442363. Epub 2016 Feb 8. PMID 26881832
- [Background] Abu Alfeilat M, Slotki I, Shavit L. Single emergency room measurement of neutrophil/lymphocyte ratio for early detection of acute kidney injury (AKI). Intern Emerg Med. 2018 Aug;13(5):717-725. doi: 10.1007/s11739-017-1715-8. Epub 2017 Jul 29. PMID 28756545
- [Background] Yilmaz H, Cakmak M, Inan O, Darcin T, Akcay A. Can neutrophil-lymphocyte ratio be independent risk factor for predicting acute kidney injury in patients with severe sepsis? Ren Fail. 2015 Mar;37(2):225-9. doi: 10.3109/0886022X.2014.982477. Epub 2014 Nov 14. PMID 25394529
- [Background] Pereira M, Rodrigues N, Godinho I, Gameiro J, Neves M, Gouveia J, Costa E Silva Z, Lopes JA. Acute kidney injury in patients with severe sepsis or septic shock: a comparison between the 'Risk, Injury, Failure, Loss of kidney function, End-stage kidney disease' (RIFLE), Acute Kidney Injury Network (AKIN) and Kidney Disease: Improving Global Outcomes (KDIGO) classifications. Clin Kidney J. 2017 Jun;10(3):332-340. doi: 10.1093/ckj/sfw107. Epub 2016 Dec 13. PMID 28616211